CLINICAL TRIAL: NCT06498648
Title: Phase I/II Study to Evaluate the Feasibility and Efficacy of Sequential Abemaciclib and Gemcitabine Treatment in Patients With Retinoblastoma (Rb)+ Sarcomas
Brief Title: Testing the Addition of an Anti-cancer Drug, Abemaciclib, to the Usual Chemotherapy Treatment (Gemcitabine) for Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-05665; NCI-2024-05665 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10657 (Other: University of Texas MD Anderson Cancer Center LAO); 10657 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Dedifferentiated Liposarcoma; Advanced Leiomyosarcoma; Advanced Soft Tissue Sarcoma; Metastatic Dedifferentiated Liposarcoma; Metastatic Leiomyosarcoma; Metastatic Soft Tissue Sarcoma; Stage III Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IV Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8
MeSH Terms: conditions — Liposarcoma; Leiomyosarcoma; Sarcoma | interventions — abemaciclib; Biopsy; Specimen Handling; Docetaxel; alovudine; Gemcitabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 2 Arm A (abemaciclib, gemcitabine) (Experimental): Patients receive abemaciclib PO BID and gemcitabine IV on the schedule determined in phase 1 of the trial. Cycles repeat every 21 or 28 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity. At the time of disease progression, patients may cross over to arm B. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy on study.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Gemcitabine
- Phase 2 Arm B (gemcitabine, docetaxel) (Active Comparator): Patients receive gemcitabine IV over 90 minutes on days 1 and 8 of each cycle and docetaxel IV over 60 minutes on day 8 of each cycle. Cycles repeat every 21 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity. At the time of disease progression, patients may cross over to arm A. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy during screening and optionally on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Docetaxel; Drug: Gemcitabine
- Phase I Part A Cohort I (abemaciclib, gemcitabine) (Experimental): Patients receive abemaciclib PO BID on days 1-5 and 15-19 of each cycle and gemcitabine IV over 90 minutes on days 8 and 22 of each cycle. Cycles repeat every 28 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity. Patients may change to Phase 1 Part B treatment once the recommended schedule is determined. Patients also receive 18F-FLT IV and undergo PET/CT during screening and on study. Additionally, patients undergo blood sample collection during screening and on study.
  Interventions: Drug: Abemaciclib; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fluorothymidine F-18; Drug: Gemcitabine; Procedure: Positron Emission Tomography
- Phase I Part A Cohort II (abemaciclib, gemcitabine) (Experimental): Patients receive abemaciclib PO BID on days 1-7 and gemcitabine IV over 90 minutes on day 10 of each cycle. Cycles repeat every 21 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity. Patients may change to Phase 1 Part B treatment once the recommended schedule is determined. Patients also receive 18F-FLT IV and undergo PET/CT during screening and on study. Additionally, patients undergo blood sample collection during screening and on study.
  Interventions: Drug: Abemaciclib; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fluorothymidine F-18; Drug: Gemcitabine; Procedure: Positron Emission Tomography
- Phase I Part B (abemaciclib, gemcitabine) (Experimental): Patients receive the selected treatment schedule, Cohort 1 or Cohort 2, as above. Cycles repeat every 21 or 28 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fluorothymidine F-18; Drug: Gemcitabine; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY 2835219; LY-2835219; LY2835219; Verzenio
  Arms: Phase 2 Arm A (abemaciclib, gemcitabine); Phase I Part A Cohort I (abemaciclib, gemcitabine); Phase I Part A Cohort II (abemaciclib, gemcitabine); Phase I Part B (abemaciclib, gemcitabine)
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Phase 2 Arm A (abemaciclib, gemcitabine); Phase 2 Arm B (gemcitabine, docetaxel)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Phase I Part A Cohort I (abemaciclib, gemcitabine); Phase I Part A Cohort II (abemaciclib, gemcitabine); Phase I Part B (abemaciclib, gemcitabine)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Phase 2 Arm B (gemcitabine, docetaxel)
Other: Fluorothymidine F-18 — Given IV
  Other Names: 18F-FLT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; ALOVUDINE F-18; Fluorothymidine F 18
  Arms: Phase I Part A Cohort I (abemaciclib, gemcitabine); Phase I Part A Cohort II (abemaciclib, gemcitabine); Phase I Part B (abemaciclib, gemcitabine)
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: Phase I Part A Cohort I (abemaciclib, gemcitabine); Phase I Part A Cohort II (abemaciclib, gemcitabine); Phase I Part B (abemaciclib, gemcitabine)

SUMMARY:
This phase I/II trial tests the side effects and best dose of abemaciclib when added to gemcitabine and compares the effectiveness of that treatment to the usual treatment of gemcitabine with docetaxel for the treatment of patients with soft tissue sarcoma that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic) (phase 1) or patients with leiomyosarcoma or dedifferentiated liposarcoma (phase 2). Abemaciclib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals tumor cells to multiply. This helps slow or stop the spread of tumor cells. Gemcitabine is a chemotherapy drug that blocks the cells from making deoxyribonucleic acid and may kill tumor cells. Docetaxel is in a class of medications called taxanes. It stops cancer cells from growing and dividing and may kill them. Giving abemaciclib with gemcitabine may be safe and effective when compared to treatment with gemcitabine and docetaxel for patients with advanced or metastatic soft tissue sarcoma or leiomyosarcoma or dedifferentiated liposarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of the phase 1 part of this trial is to define the schedule of sequential abemaciclib and gemcitabine and recommended phase 2 dose (RP2D) of retinoblastoma positive (Rb[+ve]) sarcomas.

II. The primary objective of the phase 2 part of the trial is to define the progression-free survival (PFS) of sequential abemaciclib followed by gemcitabine at RP2D compared to the standard of care gemcitabine and docetaxel in advanced Rb(+ve) leiomyosarcomas and dedifferentiated liposarcomas.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity in phase 1. II. To determine cell cycle arrest and recovery with abemaciclib 200mg twice per day (BID) 5 to 7 days by blood thymidine kinase activity (Tka).

III. To assess the toxicity profile of the sequential abemaciclib followed by gemcitabine treatment using Common Terminology Criteria for Adverse Events (CTCAE) version 5 in phase 1 & phase 2.

IV. To determine the preliminary objective response rate (ORR) by Response Criteria in Solid Tumors (RECIST)1.1 in phase 1.

V. To compare overall survival (OS) of sequential abemaciclib followed by gemcitabine at RP2D to the standard of care gemcitabine and docetaxel in phase 2.

VI. To compare the objective response rate (ORR) at time of best response by RECIST1.1 of sequential abemaciclib followed by gemcitabine at RP2D to the standard of care gemcitabine and docetaxel in phase 2.

VII. To compare PFS and ORR after cross-over in each treatment arm. VIII. To identify mechanisms of resistance to sequential treatment through correlative studies of the cell cycle genes.

EXPLORATORY OBJECTIVE:

I. To determine cell cycle arrest and recovery with abemaciclib 200mg BID 5 to 7 days by fluorothymidine F-18 (18F-FLT) positron emission tomography (PET) and its association with blood Tka.

OUTLINE: Patients in phase 1 part A are assigned to cohort 1 or 2. Patients in phase 2 are randomized to arm A or arm B and may cross over to the alternate arm after disease progression.

PHASE 1 PART A:

COHORT I: Patients receive abemaciclib orally (PO) twice per day (BID) on days 1-5 and 15-19 of each cycle and gemcitabine intravenously (IV) over 90 minutes on days 8 and 22 of each cycle. Cycles repeat every 28 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity. Patients may change to Phase 1 Part B treatment once the recommended schedule is determined. Patients also receive 18F-FLT IV and undergo PET/computed tomography (CT) during screening and on study. Additionally, patients undergo blood sample collection during screening and on study.

COHORT II: Patients receive abemaciclib PO BID on days 1-7 and gemcitabine IV over 90 minutes on day 10 of each cycle. Cycles repeat every 21 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity. Patients may change to Phase 1 Part B treatment once the recommended schedule is determined. Patients also receive 18F-FLT IV and undergo PET/CT during screening and on study. Additionally, patients undergo blood sample collection during screening and on study.

PHASE 1 PART B: Patients receive the selected treatment schedule, Cohort 1 or Cohort 2, as above. Cycles repeat every 21 or 28 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity.

PHASE 2:

ARM A: Patients receive abemaciclib PO BID and gemcitabine IV on the schedule determined in phase 1 of the trial. Cycles repeat every 21 or 28 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity. At the time of disease progression, patients may cross over to arm B. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy during screening and optionally on study.

ARM B: Patients receive gemcitabine IV over 90 minutes on days 1 and 8 of each cycle and docetaxel IV over 60 minutes on day 8 of each cycle. Cycles repeat every 21 days for up to 2 years of total treatment in the absence of disease progression or unacceptable toxicity. At the time of disease progression, patients may cross over to arm A. Patients undergo blood sample collection throughout the study. Patients also undergo tumor biopsy during screening and optionally on study.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: Patients must have advanced/metastatic histologically confirmed soft tissue sarcoma and have received at least one prior standard systemic therapy (prior gemcitabine is allowed)
* Phase 2: Patients must have advanced/metastatic pathologically confirmed leiomyosarcoma or dedifferentiated liposarcoma for which gemcitabine and docetaxel is considered standard-of-care, patients may be systemic-treatment naïve. Prior gemcitabine is not allowed
* Patients must have presence of measurable/assessable tumor
* Patients must have intact Rb gene expression in the baseline tumor biopsy or archived tumor sample, as assessed by immunohistochemistry (at MD Anderson: clone G3- 245, BD Pharmagen, RRID:AB_385259, Clinical Laboratory Improvement Act [CLIA] certified antibody)
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of abemaciclib in combination with gemcitabine in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Absolute neutrophil count ˃ 1.2K/µL
* Hemoglobin ˃ 9.0 g/dL
* Platelets ˃ 100K/mm^3
* Glomerular filtration rate (GFR) ≥ 60 mL/min unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN), patient with Gilbert's syndrome ≤ 2.0 times ULN, or direct bilirubin within normal limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) ≤ 1.5 × institutional ULN
* Alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 1.5 × institutional ULN
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association (NYHA) Functional Classification. To be eligible for this trial, patients should be class congestive heart failure (CHF) II or better
* Patients must have a life expectancy of greater than 6 months
* Females of childbearing potential must have a negative serum pregnancy test within one week of trial enrollment and be willing to use an adequate method of contraception to avoid pregnancy throughout the trial and for up to 6 months after the last dose of drug therapy. The effects of abemaciclib on the developing human fetus are unknown. For this reason and because CDK 4/6 inhibiting agents as well as gemcitabine are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of abemaciclib administration. Abstinence is considered an effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study ranging from three weeks prior to initiation of treatment and up to 6 months after the last dose of treatment
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* Patient is capable of swallowing oral medications

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents. There must be no investigational drug use within 30 days or 5 half-lives of receiving the first dose of treatment on this treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib or gemcitabine
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because abemaciclib is a CDK4/6 inhibiting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with abemaciclib or gemcitabine, breastfeeding should be discontinued if the mother is treated with abemaciclib or gemcitabine
* Use of strong CYP34A inhibitors which cannot be discontinued by the patient prior to trial initiation. The washout period of these drugs should be 5 half-lives
* Progression on prior CDK4 inhibitor therapy
* Phase 2 only: Prior gemcitabine-based chemotherapy
* Presence of significant cardiac disease. Significant cardiac disease includes personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* Patients with interstitial lung disease (ILD)
* Patients with gastrointestinal conditions that may affect the absorption of oral medications
* Patients must not have received or be scheduled to receive radiation therapy within 7 days or less from gemcitabine administration
* Patients must not have had major surgery within 14 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-04-12 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Time course of blood thymidine kinase activity (TKa) (Phase 1 Part A) | Baseline up to 2 years
  Will be graphically evaluated: the change of blood TKa over time to facilitate a selection of regimen that has maximum decrease in blood TKa after end of abemaciclib (cell cycle arrest) and has maximum increase in blood TKa at time of gemcitabine injection. Descriptive statistics (mean, standard deviation) and graphical methods will be applied to examine the distribution of the data, error checking, and outlier identification. Since blood TKa and fluorothymidine F-18 (18F-FLT) positron emission tomography (PET) will be measured at baseline and multiple post treatment time points, if appropriate, linear mixed effect models for repeated measures analysis will be employed to assess its change over time. Appropriate transformation of the marker values will be used to satisfy the normality assumption of linear mixed effect model.
Maximum tolerated dose (Phase I Part B) | Up to 28 days
Progression free survival (PFS) (phase II) | From randomization to either disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) or death from any cause, up to 2 years
  Will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Anti-tumor activity (phase I) | Up to 2 years
Cell cycle arrest (phase I) | At 5 to 7 days
  Measured by blood TKa.
Cell cycle recovery (phase I) | At 5 to 7 days
  Measured by blood TKa.
Incidence of adverse events (phase I) | Up to 2 years
  Using Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Objective response rate (ORR) (phase I) | Up to 2 years
  By Response Criteria in Solid Tumors 1.1 with a 95% exact CI will be provided.
Overall survival (phase II) | From randomization to death, up to 2 years
  Respective point estimates will be provided along with 95% confidence interval (CI) by treatment arms and then by histologic groups within treatment arm. The hazard ratio along with 95% CI using Cox proportional hazard models will be estimated. Will be estimated using the Kaplan-Meier method.
ORR at time of best response (phase II) | Up to 2 years
  A 95% exact CI will be provided.
Incidence of adverse events (phase II) | Up to 2 years
  Assessed by CTCAE v5.
Cell cycle arrest (phase II) | At day 5-7
  Measured by blood TKa.
Cell cycle recovery (phase II) | At day 5-7
  Measured by blood TKa.
Mechanisms of resistance to sequential treatment (phase II) | Up to 2 years
PFS after crossover | From randomization to either disease progression as defined by RECIST or death from any cause, up to 2 years
  Will be estimated using the Kaplan-Meier method.
ORR after crossover | Up to 2 years
  A 95% exact CI will be provided.

OTHER OUTCOMES:
Cell cycle arrest | From baseline to gemcitabine
  By 18F-FLT PET and its associations with blood TKa.
Cell cycle recovery | From baseline to gemcitabine
  By 18F-FLT PET and its associations with blood TKa.

CONTACTS AND LOCATIONS:
Overall Officials: Elise F Nassif, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm